# Understanding Engagement Trends in Chondrosarcoma Clinical Trials: Investigating Participation Patterns Among Chondrosarcoma Patients

An Informed Consent For Patients With Chondrosarcoma in Power Clinical Trial's Observational Study

Date: September 1, 2023

Information About This Consent Document

If you are requested to complete this form, it means you may be eligible to participate in observational clinical research designed exclusively for people with chondrosarcoma. This paper is a thorough guide that reveals the study's main aims, elaborate execution strategy, and multiple ramifications, both good and potentially negative. It is critical to carefully analyze your prospective participation before making a choice, and obtaining counsel from a reputable expert can give essential insights. If any of the material in this document appears confusing or if questions arise, please know that the researcher is accessible to provide an explanation.

## The Investigative Goal

Chondrosarcoma is a bone cancer that starts in cartilage cells. Cartilage is the specialized, gristly connective tissue found in adults that gives rise to the majority of bones. Cartilage is essential to the growing process. There are several forms of cartilage present throughout the body. Chondrosarcoma is a kind of cancer that typically affects cartilage cells in the femur (thighbone), arm, pelvis, or knee. Other places (such as the ribs) may be impacted less frequently.

Clinical studies aimed especially towards chondrosarcoma play an important role in determining the safety and efficacy of new therapies for this ailment. These studies are crucial in establishing whether novel medicines outperform established choices and offer strong evidence to support their widespread adoption.

This study focuses on the experiences of people diagnosed with chondrosarcoma as they actively participate in a unique clinical trial including medicinal therapies. The major focus is on closely examining trial completion rates and voluntary withdrawal rates among these individuals.

#### Unveiling the Core of Observational Studies

By taking part in this medical trial, you will be participating in an observational study, a subset of clinical research that is painstakingly structured to gather insights via unmodified monitoring of patients while maintaining their care regimens.

Researchers will just monitor your trip, thoroughly measuring the consequences of your condition while making no changes. This particular trial design is critical in furthering our understanding of the inherent evolution of a certain medical illness and its implications for people who have been diagnosed with it. By actively participating in this observational study, you actively contribute to broadening the frontiers of medical knowledge and driving improvements in the care offered to those suffering from the same illness.

## Contrasting This Trial with Other Chondrosarcoma Clinical Studies

Understanding what makes this clinical study distinctive is critical. It operates on an observational basis, which means that your participation will not entail particular therapies or interventions. Understanding the complete range of chondrosarcoma clinical trials, including interventional studies in which patients experience several treatment regimens, is critical.

Making an educated decision regarding your possible involvement in a clinical trial necessitates an active approach that includes research and comparison of various trials. Clinicaltrials.gov and other platforms provide a wealth of information regarding <a href="mailto:chondrosarcoma research">chondrosarcoma research</a>. Furthermore, Power's dedicated web hub offers a complete listing of ongoing <a href="mailto:chondrosarcoma clinical trials">chondrosarcoma clinical trials</a> that are actively recruiting volunteers.

You empower yourself to confidently design your participation decision by completing rigorous research and getting a full awareness of various clinical trial types.

#### Active Engagement in Clinical Trial Surveys

We extend a sincere invitation for you to actively share your experiences within the scope of this observational clinical investigation. This initiative requires you to complete surveys every two weeks, which will take roughly 20-30 minutes of your valuable time. Furthermore, we are fully prepared to arrange check-in calls at quarterly intervals, a commitment that will last as long as your participation in the study continues.

It is critical to emphasize that your participation in the survey portion of the trial is fully optional, as this is of the utmost significance. It is totally up to you whether you answer certain questions or finish the full questionnaire. Furthermore, you have the option to end your participation in the trial at any time. Recognizing that the choice to participate in a clinical research is deeply personal, our unchanging commitment is to provide the necessary assistance. Your privacy and comfort remain top priority, and we are committed to respecting and assisting you in making decisions throughout the course of the trial.

## Protecting the Privacy of Your Answers

Keeping your information as private as possible over the length of this clinical research is a top priority. To maintain your anonymity, please avoid including any personal or identifiable information in your questionnaire replies. The committed research team is relentless in their dedication to improving the protection of your privacy. However, you should be aware that some legal situations may develop that require the sharing of your data.

# Anticipated Advantages

While immediate benefits may not be apparent for people taking part in this observational clinical research, their participation has the potential to spread its impacts to others. The pool of data gathered from participants will be used to improve future recruitment tactics for chondrosarcoma patients, perhaps opening up new possibilities for medical study. Individuals who participate in this clinical trial have the potential to

effect dramatic change in the field of medical research, perhaps redefining the route for future chondrosarcoma sufferers.

#### **Anticipated Hazards**

Despite the extraordinary advances made possible by clinical trials, it is critical to recognize the potential health hazards that participants may face, particularly in studies testing novel therapies.

Nonetheless, our observational clinical research takes a different approach, purposefully reducing these risks by not exposing participants to novel therapies. Rather, our primary focus is on thorough monitoring and result measurement in order to avoid any unnecessary health hazards from appearing.

## **Exploring Inclusiveness in Clinical Trials**

For individuals with a strong desire to dig into the complex world of clinical trial representation, an assortment of online tools awaits your active participation.

Whether your goal is to fathom the complexities of the obstacles and possibilities associated with clinical trial diversity or to foster better knowledge, the following sources can provide insightful guidance:

Hayden, Gregory F. "Acute suppurative otitis media in children: diversity of clinical diagnostic criteria." *Clinical pediatrics* 20, no. 2 (1981): 99-104.

Farb, Andrew, Charles J. Viviano, and Michelle E. Tarver. "Diversity in Clinical Trial Enrollment and Reporting—Where We Are and the Road Ahead." *JAMA cardiology* (2023).

# Confirmation of Voluntary Agreement

I hereby certify that I have spent sufficient time comprehending and digesting the contents of the informed consent form, either via independent research or with the assistance of a trusted individual who has expressed its substance to me. All of my concerns and worries have been thoroughly handled to my entire satisfaction.

I am fully aware that my participation in this study is the product of my personal decision, and I have the only right to withdraw my consent without any requirement to offer justification or make financial commitments. I have been specifically told that a copy of this informed consent form would be supplied for my own records.

After carefully considering and evaluating all of the material offered to me, I hereby extend my permission to participate in this study, signifying my informed and self-governing decision.

| Printed Name of Participant |
|-----------------------------|
| · |
| Participant Signature |
| Date |

## Confirmation by Informed Consent Facilitator

I can certainly state that I had a full conversation with the participant, meticulously unraveling the complexities encompassed in this written paper. The goal was to ensure that the participant understood the trial's general aims, methodology, potential risks and benefits, and other critical components inherent to the chondrosarcoma clinical trial.

The participant was given ample opportunity, which encouraged the formation of questions and facilitated the explanation of concerns or misconceptions. It is critical to emphasize that the participants' participation in this study is the product of their voluntary decision, and they have the unrestricted right to withdraw at any time, for any reason, without incurring any financial responsibilities.

Following the participant's assent, they were given a meticulously kept replica of this written document, which functioned as a repository for their particular records.

| Printed Name of Person Taking Consent |
|---------------------------------------|
| Signature of Person Taking Consent |
| <br>Date |